CLINICAL TRIAL: NCT05839899
Title: Mifepristone and Misoprostol for Undesired Pregnancy of Unknown Location: A Randomized Pilot Study of Misoprostol Dosing
Brief Title: Mifepristone and Misoprostol for Undesired Pregnancy of Unknown Location
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Planned Parenthood League of Massachusetts (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023P000467
Record Dates: First submitted 2023-04-04; First posted 2023-05-03 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Abortion
MeSH Terms: interventions — Mifepristone; Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Mifepristone plus Single dose misoprostol (Active Comparator): Participant will take mifepristone, then one dose of misoprostol at home to pass the pregnancy (current routine abortion care).
  Interventions: Drug: Mifepristone plus one dose Misoprostol
- Mifepristone plus two doses misoprostol (Experimental): Participant will take mifepristone, then at home will take two doses of misoprostol 4 hours apart to pass the pregnancy.
  Interventions: Drug: Mifepristone plus two doses Misoprostol

INTERVENTIONS:
Drug: Mifepristone plus one dose Misoprostol — Mifepristone 200mg PO, then 800 mcg of misoprostol 24-30 hours later
  Arms: Mifepristone plus Single dose misoprostol
Drug: Mifepristone plus two doses Misoprostol — Mifepristone 200mg PO, then 800 mcg misoprostol 24-30 hours later, then another 800 mcg misoprostol 4 hours after that
  Arms: Mifepristone plus two doses misoprostol

SUMMARY:
Patients who seek medication abortion early in pregnancy may have an ultrasound that does not show a pregnancy in the uterus. This is known as a "pregnancy of unknown location". These patients most likely have a pregnancy in the uterus that is too early to be seen on ultrasound, but it is possible that the pregnancy is not seen inside the uterus because it is outside of the uterus, known as an ectopic pregnancy. Patients with ectopic pregnancies are at risk for serious complications, and the medications used for medication abortion may not end an ectopic pregnancy.

Currently, at Planned Parenthood League of Massachusetts (PPLM), patients seeking medication abortion, including some patients with a pregnancy of unknown location, are given mifepristone to begin the medication abortion at the clinic and then one dose of misoprostol to take at home to cause the pregnancy to pass. However, research suggests that a second dose of misoprostol leads to a higher rate of completed abortion for certain patients.

This research is being conducted to learn if two doses of the at-home misoprostol during the medication abortion process leads to a higher rate of completed abortion for patients with pregnancy of unknown location. In this study, all participants will receive mifepristone as they normally would. Then, participants will be randomly assigned to receive either one dose of misoprostol or two doses of misoprostol.

ELIGIBILITY:
Inclusion Criteria:

* Positive urine or serum hCG test
* No evidence of gestational sac on transvaginal ultrasound
* No evidence of ectopic pregnancy on transvaginal ultrasound
* Desire for same-day start medication abortion as method of pregnancy termination
* Eligible for same-day-start medication abortion based on PPLM clinical guidelines at the time of enrollment
* English-speaking

Exclusion Criteria:

* Ineligible for medication abortion at PPLM based on current PPLM clinical guidelines at the time of enrollment

  o PPLM clinical guidelines for medication abortion currently exclude those with chronic adrenal failure, concurrent long-term corticosteroid use, hemorrhagic disorders or concurrent anti-coagulation, porphyria, allergies to mifepristone or misoprostol, or an IUD in place.
* Ineligible for same-day-start medication abortion with PUL based on PPLM clinical guidelines and clinician assessment at the time of enrollment

  o PPLM clinical guidelines for initiating medication abortion with PUL currently exclude those with major ectopic risk factors (IUD in situ, prior ectopic, history of tubal surgery) or symptoms concerning for ectopic (i.e. pain, bleeding) per clinician discretion.
* Age less than 18 years old
* Prior participation in this study
* Anticipated inability to adhere to follow up protocol or complete the survey
* Unable to give informed consent or to complete all study procedures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment rates, to determine feasibility of recruitment | 1 year
  Feasibility of recruitment will be assessed by the recruitment and refusal rates. The recruitment rate will be calculated by dividing the total number of participants recruited by the number of months spent for recruitment.
Acceptability of second dose of misoprostol | 1 month per subject, 1 year for all subjects
  Acceptability of this regimen will be assessed by measuring how often patients assigned to the treatment arm actually take the second dose of misoprostol. If 13 or more patients in the double-miso group (>50%) do not take the second dose, this will be considered unacceptable.
Refusal rates, to determine feasibility of recruitment | 1 year
  Feasibility recruitment will be assessed by the recruitment and refusal rates. The refusal rate will be calculated by dividing the total number of participants recruited by the number of patients approached for study participation..

CONTACTS AND LOCATIONS:
Locations (1):
- Planned Parenthood League of Massachusetts, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available to other researchers